CLINICAL TRIAL: NCT01966744
Title: Self-Management Assistance for Recommended Treatment (SMART) Portal
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: SMART
Record Dates: First submitted 2013-10-04; First posted 2013-10-22 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; Inflammatory Bowel Disease
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Clinicians/Nurses: Clinicians and nurses who treat patients diagnosed with IBD will be recruited to interact with and use the SMART portal to provide feedback on optimization.
- Patients: Patients age 11-18 years diagnosed with IBD will be recruited to interact with and use the SMART portal to provide feedback on optimization.
- Caregivers: Caregivers of patients diagnosed with IBD will be recruited to interact with and use the SMART portal to provide feedback on optimization.

SUMMARY:
The purpose of the study is to develop, evaluate, and optimize an interactive website (the SMART portal). The SMART portal will use IBD-specific and general assessments and interventions to reduce the burden of common barriers to treatment adherence and enhance self-management skills. This study aims to build and revise the SMART portal according to feedback and testing from participants.

DETAILED DESCRIPTION:
The study consists of three phases for development and evaluation of the SMART portal. Phase 1 is the development of online assessments and intervention components. There will be no participant interaction with the portal during Phase 1. Phase 2 will consist of one, individual interview with patients, caregivers, and clinicians/nurses to interact with a portal prototype and provide feedback. Phase 3 will contain an open trial for patients and caregivers with baseline, 2-6 months interacting with the portal and progressing through applicable intervention components, and post-treatment. Patient test data will also be loaded into the portal during Phase 3 for clinicians/nurses to interact with for 2-6 months. Feedback from all users will be collected at post-treatment for optimization of the portal.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with Crohn's disease, ulcerative colitis, or indeterminate colitis (collectively known as IBD)
* Patient between 11 and 18 years of age
* Patient prescribed at least one oral medication used to treat IBD
* Access to the internet whether public (example, library) or private (example, home, personal)
* English fluency for patient, caregiver, and clinician/nurse
* Clinician/nurse currently providing medical treatment to patients diagnosed with IBD through the IBD Center at Cincinnati Children's Hospital Medical Center

Exclusion Criteria:

* Diagnosis of pervasive developmental disorder in patient or caregiver
* Diagnosis of serious mental illness (example, schizophrenia) in patient or caregiver

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients, caregivers, clinicians, and nurses will be recruited from the IBD clinic at Cincinnati Children's Hospital Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Medication adherence | Phase 3 - Approximately 2-6 months, depending upon progression through portal components
  Medication adherence will be measured by pill count data provided by patients or caregivers at baseline and post-treatment during Phase 3. Phase 3 will start approximately in October 2014 and continue through March 2015.

SECONDARY OUTCOMES:
Disease severity | Phase 3 - Approximately 2-6 months, depending upon progression through portal components
  Disease severity will be measured at baseline, post-treatment, and periodically throughout the intervention as the patient logs in to view intervention materials during Phase 3. The portal will prompt the patient to complete disease severity questions throughout the intervention, but it will be dependent upon the patient actually logging into the system. Therefore, exact time points during treatment are unknown. The Pediatric Ulcerative Colitis Activity Index (PUCAI) will be used to measure disease severity for patients diagnosed with ulcerative colitis and indeterminate colitis, and the Partial Harvey Bradshaw (PHBI) will be used for patients diagnosed with Crohn's disease. Phase 3 will start approximately in October 2014 and continue through March 2015.
Health-related quality of life | Phase 3 - Approximately 2-6 months, depending upon progression through portal components
  The IMPACT-III will be used during baseline and post-treatment in Phase 3 to measure quality of life in patients. Phase 3 will start approximately in October 2014 and continue through March 2015.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Denson, M.D., Study Chair — Children's Hospital Medical Center, Cincinnati; James Peugh, Ph.D., Study Chair — Children's Hospital Medical Center, Cincinnati; Korey Hood, Ph.D., Study Chair — University of California, San Francisco; Lee Ritterband, Ph.D., Study Chair — BeHealth Solutions, LLC.
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - BeHealth Solutions, LLC, Charlottesville, Virginia

REFERENCES:
- [Derived] Hommel KA, Ramsey RR, Gray WN, Denson LA. Digital Therapeutic Self-Management Intervention in Adolescents With Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2023 Jan 1;76(1):38-42. doi: 10.1097/MPG.0000000000003623. Epub 2022 Sep 20. PMID 36123761